CLINICAL TRIAL: NCT01873690
Title: A Randomized Controlled Trial Assessing the Efficacy of Antimicrobial Prophylaxis for Extracorporeal Shock Wave Lithotripsy on Reducing Urinary Tract Infection
Brief Title: Efficacy of Antimicrobial Prophylaxis for Shock Wave Lithotripsy (SWL) on Reducing Urinary Tract Infection (UTI)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to the low recruitment rate and the large number lost to follow-up
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Hassan Razvi, Principle Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 103696
Record Dates: First submitted 2013-06-03; First posted 2013-06-10 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Urolithiasis
Keywords: Antibiotics; Shock Wave Lithotripsy; Urinary Tract Infection
MeSH Terms: conditions — Urolithiasis; Urinary Tract Infections | interventions — Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Ciprofloxacin (Active Comparator): Ciprofloxacin
  Interventions: Drug: Ciprofloxacin

INTERVENTIONS:
Drug: Ciprofloxacin — Once, 400 mg IV
  Other Names: Ciprofloxacin Hydrochloride
  Arms: Ciprofloxacin
Drug: Placebo — 5% Dextrose in water
  Arms: Placebo

SUMMARY:
The purpose of this research study is to test whether administering one dose of an antibiotic before a routine shock wave lithotripsy procedure is more effective at avoiding any urinary infections compared to not taking an antibiotic. This is an important topic to study because urinary tract infections are one of the most common complications after this procedure and there is no clear standard of care regarding the use of pre-procedure antibiotics. Our study results will benefit future patients either by decreasing the rate of infections or decreasing the use of unnecessary antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for SWL at St. Joseph's Hospital;
* 18 years of age or older;
* Willing and able to complete Questionnaires;
* Willing to submit urine sample for analysis at Day 7;
* Able to read and speak English.

Exclusion Criteria:

* Pre-SWL urine analysis positive for nitrites or urine culture reveals >105 CFU/ml of bacteria (positive urine culture);
* Taking antibiotics for UTI or other cause;
* Requires an antibiotic post SWL;
* Suspected struvite stone (based on previous stone analysis, or partial staghorn);
* Presence of nephrostomy tube;
* Requiring cystoscopy on the day of SWL;
* Requiring ureteral stent on the day of SWL;
* Presence of indwelling urinary catheter or on regular clean intermittent catheterization (CIC);
* Presence of urinary diversion (ie: ileal conduit);
* Any history of urosepsis;
* Known allergic reaction to ciprofloxacin/quinolones;
* Patient known to be pregnant;
* Previous randomization in this trial;
* In the opinion of the urologist, it is not in the patient's best interest to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2013-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Impact of antibiotic prophylaxis on the rate of urinary tract infection | Post SWL Day 7
  Our primary outcome will be a composite endpoint comprised of: Positive post-SWL urine culture (≥ 105 colony forming units / millilitre (CFU/ml), symptoms of cystitis (defined as new onset burning sensation or pain with voiding, frequency, urgency), or pyelonephritis or urosepsis (hospital admission with fever ≥38.5 C).

SECONDARY OUTCOMES:
Bacteriuria post-SWL (≥105 cfu/ml) | 7-14 days
Symptoms of cystitis (new onset burning sensation or pain with voiding, frequency, urgency) | 7-14 days
Pyelonephritis or urosepsis (hospital admission with fever ≥38.5C) | 7-14 days
Change in Urinary Symptom Score(reported as positive or negative integer) | 7 - 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Razvi, MD, FRCSC, Principal Investigator — Western University & Lawson Research Institute
Locations (1):
- St. Joseph's Hospital, St. Joseph's Health Care London, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No